CLINICAL TRIAL: NCT05656677
Title: Pain Responses in Preterm Infants and Parental Stress Over Repeated Painful Procedures: a Randomized Pilot Trial.
Brief Title: Parental Involvement in Pain Reducing Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 079/13
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Procedural Pain; Preterm Infants; Parents
Keywords: pain; stress; preterm infants; parents
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: A three-arm pilot study using mixed methods of data collection (questionnaires, SCA, interviews) was designed to test the feasibility of the intervention encompassing parents' active and passive involvement in procedural pain management of extremely and preterm infants hospitalised at a neonatal intensive care unit (NICU).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The six NICU nurses involved were blinded to the purpose of the study, whereas the clinical nurse specialist (CNS) was not. Always three members of this research team conducted the pain assessment during the facilitated tucking or the observing by the parents. The other three members of the research team focused on the nurses' group.
  The CNS or the neonatologist provided information about the study to the parents, without stating its specific aim, instead referring in principle to the increased involvement of parents in pain management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two nurses executing facilitated tucking (FT) (No Intervention): Usual care
- One parent watching passively (Active Comparator): One parent watching passively the 2 nurses executing FT
  Interventions: Behavioral: Passive parental involvement
- One parent actively involved (Active Comparator): One parent actively executing FT
  Interventions: Radiation: Active parental involvement

INTERVENTIONS:
Behavioral: Passive parental involvement — One parent watching a procedural painful intervention, two nurses executing facilitated tucking
  Arms: One parent watching passively
Radiation: Active parental involvement — One parent watching a procedural painful intervention and at the same time executing facilitated tucking
  Arms: One parent actively involved

SUMMARY:
This pilot study was conceptualised to determine the feasibility of involving parents via facilitated tucking or observing during painful procedures and to measure change in parental stress and infant pain. An additional purpose of this pilot study was to determine the size of the cohort of preterm infants needed for a larger trial, the time, and resources required for recruitment and data collection.

DETAILED DESCRIPTION:
Objectives

In this pilot study, the aims were to determine the feasibility of whether pain behaviour in extremely and very preterm infants and perceived parental stress change when parents are involved in pain reducing measures, either actively, performing facilitated tucking or passively, observing the intervention, in comparison to the involvement of nurses only. In addition, the infant's pain reactivity and parental stress over three time points of measurement was of interest.

Methods

Extremely and very preterm infants in need of subcutaneous erythropoietin were randomly assigned to the two intervention groups. The intervention encompassed that one parent of each infant was involved during the painful procedure: Either parents executed facilitated tucking themselves or stood by, observing the procedure. Usual care involved that nurse executed facilitated tucking. All infants received 0.5ml of 30% oral glucose solution via cotton swab before the painful procedure. Infant pain was observed with the Bernese Pain Scale for Neonates (BPSN) and measured with the skin conductance algesimeter (SCA) before, during, and after the procedure. Parents' stress levels were measured before and after the painful procedure on the infant, using the Current Strain Short Questionnaire (CSSQ).

Feasibility of a subsequent trial was determined by assessing recruitment, measurement and active parental involvement. Quantitative data collection methods (i.e., questionnaires, algesimeter) were employed to determine the number of participants for a larger trial and measurement adequacy. Qualitative data (interviews) was employed to determine parents' perspectives of their involvement.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born at the NICU concerned
* Born between 24 0/7- 32 0/7 weeks of gestation, birthweight (bw) <1250g
* Infant in need of s.c. erythropoietin
* Parents fluently speaking and writing in German
* Written informed consent by parents

Exclusion Criteria:

* Premature infant with an umbilical artery pH measurement <7.00 or asphyxia
* Premature infant with life threatening malformations of the central nervous system
* Premature infant with intracranial haemorrhage (even if not present at the start of the study)
* Premature infant with any surgical intervention
* Parents with substance abuse (i.e., methadone, heroin, etc.), as mentioned in the electronic patient documentation (EPD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The main objective of this pilot study was to determine the feasibility of a larger, appropriately powered study | 1 year
  Feasibility assessment included recruitment rate (dependent on resources and in-/exclusion criteria)
Percentage of questionnaire completion | 1 year
  * Check percentage of questionnaires completed and withdrawals
  * Interview parents about the feasibility of participating three times
The pain and stress measurement over three time points were reviewed for feasibility | 1 year
  -The research team was also interviewed about acceptance, applicability and feasibility of the validated BPSN, the SCA over three time points
The active parental involvement over three time points were reviewed for feasibility | 1 year
  In semi-structured interviews, parents were asked about performing facilitated tucking or standing by as observers, acceptance, applicability and feasibility of the CSSQ and measurement over three time-points
  -The research team was also interviewed about active parental involvement

SECONDARY OUTCOMES:
The secondary interest of the study was to test for significant differences in parental stress between the two intervention and control group at three measurement points as well as infant pain. | 1 year
  To determine infant pain, two research team nurses observed the infant by using the Bernese Pain Scale for Neonates (BPSN) in real time before (2-3 minutes), during and (2-3 and 10 minutes) after the s.c. injection. The two nurses independently assessed the physiological and behavioural pain items [(18)]. The BPSN is a multidimensional tool in German and has shown satisfactory psychometric properties among preterm and term infants (validity: r = 0.75; reliability: α=0.8) [(18)].
  Skin Conductance Algesimeter (SCA) was installed before the s.c. injection until the last BPSN measurement. An electrocardiogram electrode (ECG) was placed on the sole of the foot to the left and right of the ankle of the preterm infant. An initial baseline was obtained. Subsequently, SCA pain measurement was continuous.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Zwakhalen, Prof. Dr., Study Chair — Fac. Health, Medicine and Life Sciences, Health Services Research CAPHRI - University of Maastricht
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data collection of pain assessment
Supporting Information: Study Protocol
Time Frame: 1year
Access Criteria: Personal request